CLINICAL TRIAL: NCT06527612
Title: The Effect of Exercise Training on Quality of Life and Disease Progression in Fibrosing Interstitial Lung Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, esra pehlivan, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FILD_Progression
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Fibrosis, Pulmonary; Pulmonary Rehabilitation
Keywords: ILD; fibrosis; exercise; pulmonary rehabilitation
MeSH Terms: conditions — Pulmonary Fibrosis; Fibrosis; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): In addition to standard medical treatment, the EGr will undergo an exercise program. The initial exercise training will be conducted in the hospital, followed by online exercise sessions via video conferencing three times a week during the first week. From the second week onwards, they will be asked to perform their exercises at home three times a week using provided exercise videos and will be monitored for one year. Compliance with the exercise regimen will be assessed through a weekly survey shared in a WhatsApp group established for the exercise group patients.
  Interventions: Other: Pulmonary rehabilitation exercise programme
- Control group (No Intervention): Patients in the CGr will receive an information brochure containing medical treatment and physical activity recommendations.

INTERVENTIONS:
Other: Pulmonary rehabilitation exercise programme — In addition to standard medical treatment, the EGr will undergo an exercise program. The initial exercise training will be conducted in the hospital, followed by online exercise sessions via video conferencing three times a week during the first week. From the second week onwards, they will be asked to perform their exercises at home three times a week using provided exercise videos and will be monitored for one year. Compliance with the exercise regimen will be assessed through a weekly survey shared in a WhatsApp group established for the exercise group patients.
  Arms: Exercise Group

SUMMARY:
In this study, the progression of the disease and changes in quality of life will be examined over a 1-year follow-up period in groups of patients with Fibrosing Interstitial Lung Disease who either participated in or did not participate in a pulmonary rehabilitation program. After the initial evaluation, the patients will be randomized into two groups: one serving as the control group and the other as the pulmonary rehabilitation exercise group.

DETAILED DESCRIPTION:
Patients diagnosed with fibrosing lung disease by a pulmonology specialist at Yedikule Chest Diseases and Thoracic Surgery Training and Research Hospital will be included in the study. Those meeting the inclusion criteria will be randomized into two groups: the Exercise Group (EGr) and the Control Group (CGr). After the initial evaluation, patients will be assessed at 3, 6, and 12 months. They will be called back to the hospital for follow-up evaluations. In addition to standard medical treatment, the EGr will undergo an exercise program. The initial exercise training will be conducted in the hospital, followed by online exercise sessions via video conferencing three times a week during the first week. From the second week onwards, they will be asked to perform their exercises at home three times a week using provided exercise videos and will be monitored for one year. Compliance with the exercise regimen will be assessed through a weekly survey shared in a WhatsApp group established for the exercise group patients. Patients in the CGr will receive an information brochure containing medical treatment and physical activity recommendations

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-75 years
* Diagnosed with fibrosing interstitial lung disease according to the clinical diagnostic criteria of the American Thoracic Society and European Respiratory Society (ATS-ERS)
* Presence of dyspnea on exertion
* Stable clinical condition at the time of inclusion without infection or exacerbation in the previous 4 weeks
* Proficiency in using a smartphone

Exclusion Criteria:

* Severe comorbid diseases, unstable coronary artery disease, collagen vascular diseases, or requiring high-flow oxygen therapy (> 3-4 L/min)
* History of exertional syncope or any comorbidity that prevents exercise training (such as severe orthopedic or neurological deficits or unstable heart disease)
* Participation in a pulmonary rehabilitation program within the last 12 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-07-29 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Saint George Quality of life questionnaire | Baseline, at 3rd, 6th and 12th months after the intervention
  Saint George Respiratory Questionaire (SGRQ) score: The SGRQ ranges from 0 (no impairment of quality of life) to 100 (highest impairment of quality of life).
Forced vital capacity | Baseline, at 3rd, 6th and 12th months after the intervention
  It will perform by using the Pony Fx spirometry device, and according to the American Thoracic Society (ATS) guidelines.
Diffusing Capacity of the Lungs for Carbon Monoxide | Baseline, at 3rd, 6th and 12th months after the intervention
  Diffusing Capacity of the Lungs for Carbon Monoxide (DLCO) measurement will be conducted as part of the study to assess the lung function of participants. This test evaluates how well gases such as oxygen are transferred from the lungs to the blood.
Peripheral oxygen saturation | Baseline, at 3rd, 6th and 12th months after the intervention
  Peripheral oxygen saturation (SpO2) will be measured to assess the oxygen level in the blood. This non-invasive test provides an indication of how well oxygen is being transported to the extremities of the body, which is essential for evaluating respiratory function.

SECONDARY OUTCOMES:
Six minute walking test | Baseline, at 3rd, 6th and 12th months after the intervention
  The 6-minute walking test will conduct in a 30-meter corridor in line with American Thoracic Society (ATS) guidelines. Participants will ask to walk as far as they can. Prior to and following the test, oxygen saturation, heart rate and Borg fatigue rating will measure, and the walking distance will record.
Peripheral muscle strength | Baseline, at 3rd, 6th and 12th months after the intervention
  Peripheral muscle strength will be assessed using a digital dynamometer. This device measures the maximum force exerted by muscles in various extremities, providing quantitative data on muscle strength. The measurements will help evaluate the participants' muscle function and overall physical condition.
Modified Medical Research Council Dyspnea Score | Baseline, at 3rd, 6th and 12th months after the intervention
  Modified Medical Council Dyspnea score will rate the sensation of dyspnea as the person perceives it.The severity of dyspnea is rated on a scale of 0 to 4."0 point" means no dyspnea perception and "4point" means severe dyspnea perception.
Leicester cough questionnaire | Baseline, at 3rd, 6th and 12th months after the intervention
  The Leicester Cough Questionnaire (LCQ) consists of 19 items divided into three domains: physical, psychological, and social. Each item is scored on a 7-point Likert scale, where 1 indicates the greatest impairment and 7 indicates no impairment. The scores from each domain are summed to provide a total score, with higher scores indicating a better quality of life and fewer symptoms related to chronic cough. The maximum total score is 21, reflecting the best possible quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Esra Pehli̇van, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No